CLINICAL TRIAL: NCT04317261
Title: Role of Novel Urinary Genomic and Metablomic Markers in Diagnosis of Bladder Cancer in Patients With Hematuria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amr Abdel-Lateif El-Sawy, Principal Investigator, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AE 4320
Record Dates: First submitted 2020-03-04; First posted 2020-03-23 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Hematuria; Bladder Cancer
Keywords: Hematuria; Bladder cancer; Biomarkers; mRNA; Cytology; metabolomics
MeSH Terms: conditions — Hematuria; Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hematuria patients (Experimental)
  Interventions: Diagnostic Test: Xpert Bladder Cancer Monitor (Xpert Monitor) test and assay of urinary metabolomics (gene expression of CRAT and SLC)

INTERVENTIONS:
Diagnostic Test: Xpert Bladder Cancer Monitor (Xpert Monitor) test and assay of urinary metabolomics (gene expression of CRAT and SLC) — Urine sample is evaluated for RNA and urinary metabolites

SUMMARY:
Our goal is to develop a noninvasive, fast and simple assay to detect BCa on the GeneXpert system and metablomic genes.

DETAILED DESCRIPTION:
The Xpert BCa monitor is a novel mRNA-based urine test that measures five mRNA targets (ABL1, ANXA10, UPK1B, CRH, and IGF2) in urine sample by real time RT-PCR. Previous studies had investigated the feasibility and diagnostic performance characteristics of Xpert monitor for surveillance of NMIBC patients (12, 13). It demonstrated a high SN and NPV in relation to urine cytology.

On the other hand, metabolic dysfunction has been implicated in a wide variety of human diseases including BC (14). Growth and division of tumor cells are associated with an increase in the activity of a variety of metabolic pathways. Significant alterations in the carnitine-acylcarnitine metabolic pathways were detected in urine speci¬mens from BC patients compared to those of healthy controls (15). The expression of six genes involved in the carnitine-acylcarni¬tine metabolic pathway (CPT1A, CPT1B, CPT1C, CPT2, SLC25A20, and CRAT) was assessed by Won and colleagues. CRAT and SLC25A20 were found to be significantly down regulated in BC patients (16).

In this context, we aimed in the current study at prospective assessment of diagnostic performance characteristics of Xpert Bladder Cancer Monitor (Xpert Monitor) test and urinary metabolomics (urinary metabolites of tissue mRNA genes expression CRAT and SLC 25A20) for bladder cancer detection in patients with hematuria.

ELIGIBILITY:
Inclusion Criteria:

* Patients with gross or persistent microscopic hematuria with irritative bladder symptoms

Exclusion Criteria:

* patients on anticoagulants
* patients with history of radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance of Xpert Bladder Cancer Monitor (Xpert Monitor) test | 1 year
  Diagnostic performance of Xpert Bladder Cancer Monitor (Xpert Monitor) test for bladder cancer detection in patients with hematuria
Diagnostic performance of assay of urinary metabolomics (gene expression of CRAT and SLC) | 1 year
  Diagnostic performance of assay of urinary metabolomics (gene expression of CRAT and SLC) for bladder cancer detection in patients with hematuria

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Undecided